CLINICAL TRIAL: NCT02058771
Title: ULTIMATE: Utilising Lifemap to Investigate Malignant Arrhythmia ThErapy
Brief Title: Utilising Lifemap to Investigate Malignant Arrhythmia Therapy
Acronym: ULTIMATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospitals, Leicester (Other)
Collaborators: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: UHL10824: ULTIMATE
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Ischemic Cardiomyopathy; Sudden Cardiac Death; Implantable Defibrillator User; Myocardial Infarction; Arrhythmias, Cardiac
Keywords: Action potential duration restitution; Ventricular arrhythmia; Sudden cardiac death; Body-surface potential mapping; Electrocardiogram
MeSH Terms: conditions — Death, Sudden, Cardiac; Myocardial Infarction; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fresh Frozen Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ischaemic cardiomyopathy: Patients with ischaemic cardiomyopathy attending for ICD implantation

SUMMARY:
It is universally recognised that current methods for risk stratification of sudden cardiac death (SCD) are limited. A novel SCD risk marker, the Regional Restitution Instability Index (R2I2), measures the degree of heterogeneity in electrical restitution using data obtained from a standard 12 lead ECG acquired during an invasive electrophysiological study.

In an ischaemic cardiomyopathy (ICM) cohort of 66 patients, an R2I2 of ≥1.03 identified subjects with a significantly higher risk of ventricular arrhythmia (VA) or death (43%) compared with those with an R2I2 <1.03 (11%) (P=0.004).

This study will use non-invasive techniques to acquire electrical restitution data: exercise and pharmacological stress, and will incorporate body surface potential mapping to develop a non-invasive and high-resolution form of R2I2. Suitable patients will be recruited into a prospective, observational study.

HYPOTHESES:

PRIMARY:

1. R2I2 is predictive of ventricular arrhythmia (VA) / SCD in patients with ICM.
2. The exercise stress protocol will create a dynamic range of heart rates that allows ECG quantification of electrical restitution heterogeneity that correlates with invasive R2I2 and is predictive of VA/SCD. The pharmacological stress protocol will create a dynamic range of heart rates that allows ECG based quantification of electrical restitution heterogeneity that correlates with invasive R2I2 and is predictive of VA/SCD.

SECONDARY:

1. A high-resolution electrical map acquired using body surface potential mapping will correlate with R2I2 and these data can be included in the R2I2 calculation to improve its prediction of SCD/VA.
2. Serial measurement of R2I2 will produce consistent values.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* History of ischaemic cardiomyopathy

Exclusion Criteria:

* Unable to give informed consent
* <28 days since cardiac surgery or acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ischaemic cardiomyopathy attending for ICD implantation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Ventricular arrhythmia/Sudden cardiac death | 18 months

SECONDARY OUTCOMES:
Syncope | 18 months
All cause mortality | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: G. Andre Ng, MBChB, PhD, Principal Investigator — University of Leicester
Locations (1):
- NIHR Leicester Cardiovascular Biomedical Research Unit, Leicester, United Kingdom